CLINICAL TRIAL: NCT05925361
Title: Pedicled Peritoneum Vaginoplasty in Feminizing Genital Surgery; Implementation According to IDEAL Framework
Brief Title: Peritoneum Vaginoplasty; Implementation According to IDEAL Framework
Acronym: PeriVaS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, prof. dr. Mark-Bram Bouman, MD PhD, Clinical Professor in plastic surgery and Head of department of Plastic Surgery, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL80365
Record Dates: First submitted 2022-02-07; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Rokitansky Kuster Hauser Syndrome; Vaginal Neoplasms; Gender Incongruence; Vaginal Obstruction; Penoscrotal Hypoplasia
MeSH Terms: conditions — Mullerian aplasia; Vaginal Neoplasms; Gender Dysphoria

STUDY DESIGN:
Intervention Model Description: Single center prospective intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): All participants will undergo a laparoscopic single flap peritoneum vaginoplasty
  Interventions: Procedure: Laparoscopic pedicled single flap peritoneum vaginoplasty

INTERVENTIONS:
Procedure: Laparoscopic pedicled single flap peritoneum vaginoplasty — After the perineal part of the operation, in which the vaginal cavity will be dissected, a laparoscopy will be started. During laparoscopy, a single flap peritoneum will be harvested. The flap will be checked for adequate blood supply. The flap will be brought down to the (neo) vaginal cavity and sutured around a dilatator cylinder wise.

SUMMARY:
This study aims to assess if a single flap peritoneum vaginoplasty is safe and feasible.The IDEAL framework for evaluation and implementation of surgical techniques will be used. There are two patient groups who are eligible to undergo this procedure. The first group consists of transgender women who either have a shortage of penile skin (so they cannot undergo standard operation technique: penile inversion) or a stenosis of their primary neovagina. The second group consists of women who are born without a vagina or have an acquired short or absent vagina after vaginectomy or hysterectomy because of malignancy of the cervix or vagina. At the moment, standard procedure for both groups in the Amsterdam University Medical Center (UMC) is the sigmoid vaginoplasty, where a part of the bowel is used to form a vaginal cavity. This procedure is risky, because in some cases, the bowel anastomosis is defect. An other more frequent complication, is malodorous excessive discharge. Sometimes accompanied by inflammation of the diversion neovagina.

In recent years, the use of the peritoneum vaginoplasty has been described for transgender women. However, the peritoneum is either used as small flaps to deepen the vagina, or the peritoneum is pulled down, which limits the depth of the neovagina. We want to implement a different technique, where the peritoneum is harvested in a single pedicled flap, which is brought down and sutured in the cavity cylinder shaped. The risks are the same as in any laparoscopic surgery, but we suspect the risk of failure of the anastomosis is much lower, as is the chance of a temporary stoma.

DETAILED DESCRIPTION:
Vaginoplasty is the surgical (re)construction of a neo- vagina. At the moment, the standard procedure to construct a neo-vagina is a penile inversion vaginoplasty. Where the skin of the penis is used as lining of the neovagina. When there is insufficient or no penile skin available, up to now the standard procedure is to form a neovagina through a diversion of the large bowel. This entails extensive colorectal surgery with potential major morbidity. Another complication of this procedure that is more frequent, is malodorous excessive discharge due to colitis of the bowel conduit. Furthermore, ant theoretical risk of malignancy of the diversion vagina is present due to the chronic inflammations. A less morbid peritoneum 'pull down' vaginoplasty is a well-known and widely used alternative technique for cis-women who are born without a vagina. However, the technique limits the maximum achievable depth and subsequent functional outcome. By using a single pedicled peritoneum flap, it is possible to create more depth.

In recent years, the peritoneum vaginoplasty is also performed in transgender women, with reported good results. However, in these publications the peritoneum is either used as small flaps to deepen the vagina, or the peritoneum is pulled down. The investigators propose to introduce an optimized technique, based upon a single pedicled peritoneal flap, which is brought down and sutured in the vaginal cavity to form a cylinder. The perioperative risks are suspected to be substantially lower with minimal chance of bowel leakage and thereby the risk on re-interventions or a temporary stoma. Second, at long term the chance of malodorous discharge and chronic inflammation is lower, which is expected to result in improved satisfaction and sexual function.

This study aims to assess if the single flap pedicled peritoneum vaginoplasty is safe and feasible in transgender women with penoscrotal hypoplasia or obliteration of the primary neovagina and in cis-women with congenital or acquired lack of vaginal depth.

ELIGIBILITY:
Inclusion Criteria:

* Indication for vaginoplasty, with no option to use penoscrotal tissue or with shortage of penoscrotal tissue.
* Age >18
* Able to give informed consent

Exclusion Criteria:

* Contra-indication for laparoscopic surgery
* Smoking (cessation for at least 6 weeks)
* BMI 18 < or >30 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — one of two groups consists of transgender or gender diverse individuals, who desire feminizing genital surgery. So they are assigned male at birth, but identify as female or gender diverse.
Enrollment: 13 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
90 day postoperative complications. Reported by full description of the event and eventual treatment and classified according to Clavien-Dindo classification. | From start of surgery until 90 days after surgery
  Reported by full description of the event and eventual treatment and classified according to Clavien-Dindo classification.

SECONDARY OUTCOMES:
Successful technical completion of operation | From start of surgery until 90 days after
  Postoperative dimension of the neovagina of at least 12 cm, measured by a measuring dilatator.
Operation time | Intraoperative (From start of surgery up until closure of all wounds)
  Learning curve of surgeons
Blood loss | Intraoperative (From start of surgery up until closure of all wounds)
  Total estimated blood loss during operation by surgeon in ml
Length of hospital stay | From date of operation/intervention until the date of discharge or death, whichever came first, assessed up to 100 days
  The total amount of days spend in the hospital after operation up until discharge.
Sexual function | at 12 months post-operation
  Sexual function measured by the sexual function form of the genderQ
Urinary function | at 12 months post-operation
  Urinary function measured by the urinary function form of the genderQ
Post-operative pain | at 3 weeks, 3 months and 6 months post-operative
  Postoperative pain reported by patient either none-normal-or excessive
Neovaginal dimensions | at 3 weeks, 3 months and 6 months post-operative
  Postoperative dimension of the neovagina, measured by a measuring dilatator.
Clitoral sensation | at 3 weeks, 3 months and 6 months post-operative
  patient assessed outcome, either none- less- normal or hyper

CONTACTS AND LOCATIONS:
Overall Officials: Mark-Bram Bouman, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam University Medical Center, Amsterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Sluis WB, Bouman M, Meijerink W, Neefjes-Borst EA, van Bodegraven AA. Refractory diversion neovaginitis in a sigmoid-colon-derived neovagina: clinical and histopathological considerations. Frontline Gastroenterol. 2016 Jul;7(3):227-230. doi: 10.1136/flgastro-2015-100602. Epub 2015 Jun 4. PMID 28839860
- [Background] van der Sluis WB, Bouman MB, Meijerink WJHJ, Elfering L, Mullender MG, de Boer NKH, van Bodegraven AA. Diversion neovaginitis after sigmoid vaginoplasty: endoscopic and clinical characteristics. Fertil Steril. 2016 Mar;105(3):834-839.e1. doi: 10.1016/j.fertnstert.2015.11.013. Epub 2015 Nov 26. PMID 26632208
- [Background] Qin C, Luo G, Du M, Liao S, Wang C, Xu K, Tang J, Li B, Zhang J, Pan H, Ball TW, Fang Y. The clinical application of laparoscope-assisted peritoneal vaginoplasty for the treatment of congenital absence of vagina. Int J Gynaecol Obstet. 2016 Jun;133(3):320-4. doi: 10.1016/j.ijgo.2015.11.015. Epub 2016 Mar 2. PMID 27087418
- [Background] Jacoby A, Maliha S, Granieri MA, Cohen O, Dy GW, Bluebond-Langner R, Zhao LC. Robotic Davydov Peritoneal Flap Vaginoplasty for Augmentation of Vaginal Depth in Feminizing Vaginoplasty. J Urol. 2019 Jun;201(6):1171-1176. doi: 10.1097/JU.0000000000000107. PMID 30707129
- [Background] Jun MS, Gonzalez E, Zhao LC, Bluebond-Langner R. Penile Inversion Vaginoplasty with Robotically Assisted Peritoneal Flaps. Plast Reconstr Surg. 2021 Aug 1;148(2):439-442. doi: 10.1097/PRS.0000000000008198. No abstract available. PMID 34398096
- [Background] Salibian AA, Schechter LS, Kuzon WM, Bouman MB, van der Sluis WB, Zhao LC, Bluebond-Langner R. Vaginal Canal Reconstruction in Penile Inversion Vaginoplasty with Flaps, Peritoneum, or Skin Grafts: Where Is the Evidence? Plast Reconstr Surg. 2021 Apr 1;147(4):634e-643e. doi: 10.1097/PRS.0000000000007779. PMID 33776039